CLINICAL TRIAL: NCT03382340
Title: A Phase 1/2a Open-Label, Dose-Escalation/Dose-Expansion Safety, Tolerability and Pharmacokinetic Study of IMX-110 in Patients With Advanced Solid Tumors
Brief Title: IMX-110 in Patients With Advanced Solid Tumors
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Immix Biopharma Australia Pty Ltd (Industry)
Responsible Party: Sponsor
Organization: Immix Biopharma, Inc. (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IMX-110-001
Record Dates: First submitted 2017-12-15; First posted 2017-12-22 (Actual); Last update posted 2023-09-28 (Actual); Status verified 2023-09

CONDITIONS: Solid Tumor, Adult; Advanced Solid Tumors; Pancreatic Cancer; Breast Cancer; Ovarian Cancer
MeSH Terms: conditions — Pancreatic Neoplasms; Breast Neoplasms; Ovarian Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Imx-110 (Experimental)
  Interventions: Drug: Imx-110

INTERVENTIONS:
Drug: Imx-110 — a nanoparticle encapsulating a Stat3/NF-kB/poly-tyrosine kinase inhibitor and low-dose doxorubicin

SUMMARY:
Phase 1 is an open-label, multi-center dose escalation/dose expansion study designed to assess the safety, tolerability and pharmacokinetics (PK) for the recommended phase 2 dose (RP2D) of IMX-110. The RP2D will be evaluated in a further dose expansion Phase 2a study submitted.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female patients who are 18 years or older
2. Patients with confirmed advanced solid tumor as per histology, who have progressed, are refractory, or are intolerant to standard therapy appropriate for tumor type
3. Patients with an Eastern Cooperative Oncology Group (ECOG) Performance status of 0-2 (Appendix 2)
4. Patients with a life expectancy of at least 3 months
5. Patients with adequate cardiac function as measured by left ventricular ejection fraction >50%
6. Patients who meet the following laboratory requirements:

   1. Absolute neutrophil count (ANC) ≥ 1.0 x 10^9/L
   2. Hemoglobin (HGB) ≥ 90.0 g/L (patients may be transfused to achieve this HGB level)
   3. Platelet count ≥ 100 x 10^9/L
   4. Total bilirubin level ≤ 1.5 x ULN
   5. AST and ALT ≤ 2.5 x ULN (≤5 x ULN if liver metastasis present)
   6. Creatinine ≤ 1.5 x ULN (Creatinine clearance >50 mL/min/1.73 m2 for subjects with creatinine levels above institutional normal)
7. Women of childbearing potential and men must agree to use highly effective, double barrier contraception during the study and for 6 weeks following the final dose of IMX-110. Double barrier contraception is defined as a condom AND one other form of the following:

   1. Birth control pills (The Pill)
   2. Depot or injectable birth control
   3. IUD (Intrauterine Device)
   4. Birth control patch (e.g. Ortho Evra)
   5. NuvaRing®
   6. Documented evidence of surgical sterilization at least 6 months prior to the screening visit, i.e., tubal ligation or hysterectomy for women or vasectomy for men.

Male patients must not donate sperm for at least 24 weeks post-dose of the last study treatment. Male partners of female patients and female partners of male patients must also use contraception, if they are of childbearing potential.

Females of childbearing potential must have a negative serum pregnancy test at Screening and a negative urine pregnancy test on Day -1.

Rhythm methods during the study and for 6 weeks after the dose of IMX-110 will not be acceptable.

Exclusion Criteria:

1. Patients with a history of severe allergic reactions to any unknown allergens or any components of the study drug formulation.
2. Patients receiving any chemotherapy within 14 days of dosing, immunotherapy within 28 days of dosing, or biologic or hormonal therapy within 28 days of dosing for cancer treatment. Patients with prostate cancer can continue administration of Gonadotropin-releasing hormone (GnRH) agonists.
3. Subject participating in any other drug study ≤ 4 weeks (6 weeks for immunotherapy investigational agents) or 5 half-lives of the investigational product, whichever is longer, prior to study drug administration or is scheduled to receive one during the treatment or post-treatment period.
4. Patients who have reached their life time limit of DOX or who are anticipated to reach their lifetime limit (550 mg/m2) within the first 2 cycles of IMX-110 administration.
5. Patients who are expected to need surgery or benefit from other anti-cancer therapy to be initiated during the study period.
6. Patients with a history of and/or risk factors for ischemic heart disease, congestive heart failure, symptomatic bradycardia, atrioventricular (AV) block, prolonged QTcF interval (>450 msec in men and >470 msec in women and additional risk factors for QT prolongation (e.g. hyperthyroidism, electrolyte imbalance).
7. Patients who have not recovered from adverse events (AEs; ≥ CTCAE grade 2) due to prior treatment (i.e. chemotherapy, targeted therapy, radiation, or surgery) within 7 days prior to Cycle 1 Day 1, unless deemed to be irreversible, or approved by the Sponsor and Medical Monitor.
8. Females who are pregnant or lactating or intend to become pregnant before, during, or within 24 weeks after participating in this study; or intending to donate ova during such time period.
9. Patients with a known positive test for human immunodeficiency virus (HIV), hepatitis B surface antigen (HBsAg) or hepatitis C antibodies (HCV). Patients may be enrolled if they have HBV or HCV with viral load suppressed by anti-virals.
10. Any condition that, in the opinion of the investigator or sponsor, would interfere with evaluation of the investigational product.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2018-02-15 (Actual); Primary Completion 2023-10-31 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Number of participants with treatment-related adverse events assessed by CTCAE v4.03. | 28 days
Maximum tolerated dose (MTD) of IMX-110 in patients with advanced solid tumors for evaluation in Phase 2a. | 28 days
  The MTD is defined as the highest dose at which ≤ 33% of the patients treated during the 3+3 design experience a DLT and/or at least two ≥ grade 2 toxicities during the first treatment cycle, and will be used to identify the RP2D to be taken forward to Phase 2a.
Recommended Phase 2 Dose (RP2D) of IMX-110 in patients with advanced solid tumors | 28 days
  RP2D is defined as one dose level below MTD

SECONDARY OUTCOMES:
Plasma concentrations of IMX-110 | 5 days
  Plasma concentrations of IMX-110 will be measured when administered in treatment Cycle 1. Samples will be collected on the first day (pre-dose, 0.5, 1, 2, 4, 6 and 24 hours post-dose) and the 5th day of dosing (pre-dose, 0.5, 1, 2, 4 and 6 hours post-dose).
Response Rate | 8 weeks
  Objective Response Rate as determined by Response Evaluation Criteria in Solid Tumors (RECIST) criteria version 1.1.
Progression-free survival (PFS) | 5 years
  PFS is measured from the start of treatment to the time of progression or death, whichever occurs first while on the study.
Overall Survival (OS) | 5 years
  OS is defined as the time from Cycle 1 Day1 to death due to any cause.
Duration of Response (DOR) | 5 years
  DOR as determined by RECIST criteria version 1.1.

OTHER OUTCOMES:
Pharmacodynamic activity of IMX-110 with appropriate biomarkers. | Baseline and the end of Cycle 1 (each cycle is 28 days)

CONTACTS AND LOCATIONS:
Locations (2):
- Sarcoma Oncology Research Center, Santa Monica, California, United States
- St George Hospital, Sydney, New South Wales, Australia